CLINICAL TRIAL: NCT01200420
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Antiviral Activity of SPC3649 (Miravirsen) Administered to Treatment-Naïve Subjects With Chronic Hepatitis C (CHC) Infection
Brief Title: Multiple Ascending Dose Study of Miravirsen in Treatment-Naïve Chronic Hepatitis C Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPC3649-203; 2010-019057-17 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Hepatitis C
Keywords: Antisense; miR-122 antagonist; host factor; CHC
MeSH Terms: conditions — Hepatitis C | interventions — miravirsen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- miravirsen (Experimental): Dose escalation study with review of safety data following each cohort.
  Interventions: Drug: miravirsen
- saline (Placebo Comparator): Dose escalation study with review of safety data following each cohort.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: miravirsen — SC injection
  Other Names: SPC3649
  Arms: miravirsen
Drug: saline — SC injection
  Arms: saline

SUMMARY:
The main purpose of this study is to determine the safety and tolerability of multiple dosing of miravirsen in subjects infected with chronic hepatitis C.

Secondary purpose includes assessment of pharmacokinetics of miravirsen and assessment of miravirsen's effect on HCV viral titer.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-38 kg/m2
* Treatment-naïve to interferon-alpha based therapies
* HCV genotype 1
* Clinical and laboratory findings consistent with a clinical diagnosis of CHC, including:

Previous documentation of positive HCV serology (HCV antibody or HCV RNA) at least 24 weeks prior to enrollment, OR Positive HCV serology (HCV antibody or HCV RNA) with a prior remote risk factor (more than 24 weeks prior to Screening) for the acquisition of hepatitis C

* Serum HCV RNA > 75,000 IU/mL at Screening
* (North American sites only). Liver biopsy within 36 months of Day 1, indicating the absence of cirrhosis
* Screening hematology, clinical chemistries, coagulation and urinalysis are not clinically significant and the following criteria are met:
* Platelets >100,000/mm3
* Total WBC > 3000/mm3 and ANC >1500/mm3
* Hemoglobin > 11 g/dL for females and > 12 g/dL for males
* Total and direct bilirubin, WNL (except for clearly documented Gilbert's Syndrome)
* ALT < 5 x ULN
* Serum creatinine WNL and creatinine clearance as calculated by the Cockcroft-Gault formula > 80 ml/min
* Negative results on the following Screening laboratory tests: urine or serum pregnancy test (for women of childbearing potential), hepatitis B surface antigen and human immunodeficiency virus (HIV) antibody.
* For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner become pregnant) during the full course of the study. Adequate contraceptive measures include oral contraceptives (stable use for 2 or more cycles prior to Screening). IUD, Depo-Provera, Norplant System implants, bilateral tubal ligation, vasectomy, condom or diaphragm plus either contraceptive sponge, foam or jelly and abstinence.

Exclusion Criteria:

* Other known cause of liver disease except for CHC
* History or symptoms of decompensated liver disease: Child-Pugh Class B or C, including ascites, hepatic encephalopathy, esophageal variceal bleeding, fibrosis or other signs of hepatic insufficiency or portal hypertension
* History of hepatocellular carcinoma (HCC) on imaging studies or serum alpha-fetoprotein (AFP) > 50 ng/mL at Screening
* Concurrent clinically significant medical diagnosis (other than hepatitis C-related conditions) that would potentially interfere with the subjects study compliance or confound study results
* Concurrent social conditions (e.g. drugs, alcohol, transportation) which would potentially interfere with the subject's study compliance
* Clinically significant illness within 30 days preceding entry into the study
* Participated in an investigational drug study within 30 days or 5 half-lives, whichever is longer, prior to the start of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | regularly over 18 weeks
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs, 12 lead and ECG monitoring.

SECONDARY OUTCOMES:
Pharmacokinetics | continuously over 4 weeks
  Appropriate PK parameters, e.g. maximum observed plasma drug concentrations, area under the plasma concentration-time curves, the apparent terminal rate constant and corresponding half-life for miravirsen.
Miravirsen treatment effect on viral titer | regularly over 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zeuzem, MD, Principal Investigator — J.W. Goethe University Hospital, Frankfurt
Locations (7):
- Alamo Medical Research, San Antonio, Texas, United States
- J.W. Goethe University Hospital, Frankfurt, Germany
- Netherlands (2):
  - Academic Medical Center (AMC), Amsterdam
  - Erasmus MC University Hospital, Rotterdam
- Klinika Hepatologii i Nabytych Niedoborow Immunologicznych WUM, Warsaw, Poland
- Fundacion de Investigation de Diego, San Juan, Puerto Rico
- FNsP Bratislava, Nemocnica akad., Bratislava, Slovakia

REFERENCES:
- [Derived] Ottosen S, Parsley TB, Yang L, Zeh K, van Doorn LJ, van der Veer E, Raney AK, Hodges MR, Patick AK. In vitro antiviral activity and preclinical and clinical resistance profile of miravirsen, a novel anti-hepatitis C virus therapeutic targeting the human factor miR-122. Antimicrob Agents Chemother. 2015 Jan;59(1):599-608. doi: 10.1128/AAC.04220-14. Epub 2014 Nov 10. PMID 25385103
- [Derived] Janssen HL, Reesink HW, Lawitz EJ, Zeuzem S, Rodriguez-Torres M, Patel K, van der Meer AJ, Patick AK, Chen A, Zhou Y, Persson R, King BD, Kauppinen S, Levin AA, Hodges MR. Treatment of HCV infection by targeting microRNA. N Engl J Med. 2013 May 2;368(18):1685-94. doi: 10.1056/NEJMoa1209026. Epub 2013 Mar 27. PMID 23534542